CLINICAL TRIAL: NCT06848894
Title: Efficacy and Safety of Human Urinary Kallidinogenase for Acute Ischemic Stroke Patients Receiving Reperfusion Treatment
Acronym: UNITE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, yilong Wang, Executive Vice-President, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY2024-320-04
Record Dates: First submitted 2025-02-20; First posted 2025-02-27 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Acute Ischemic Stroke
Keywords: Human Urinary Kallidinogenase; Acute Ischemic Stroke; Reperfusion Treatment
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): HUK (0.15 PNA) and sodium chloride injection (100ml), once per day
  Interventions: Drug: Human urinary kallidinogenase (HUK)
- Control group (Placebo Comparator): placebo (0 PNA) and sodium chloride injection (100ml), once per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Human urinary kallidinogenase (HUK) — HUK (0.15 PNA) and sodium chloride injection (100ml), once per day
  Arms: Intervention group
Drug: Placebo — placebo (0 PNA) and sodium chloride injection (100ml), once per day
  Arms: Control group

SUMMARY:
This study aims to explore the efficacy and safety of Human Urinary Kallidinogenase for acute ischemic stroke patients receiving intravenous thrombolysis and/or endovascular treatment.

DETAILED DESCRIPTION:
Within 24 hours after symptom onset, eligible participants will be randomly assigned in a 1:1 ratio to the HUK or placebo group, receiving adjunctive HUK or placebo treatment alongside standard intravenous thrombolysis and/or endovascular treatment. All participants will be recommended to continuously inject drugs or placebo for 10 to 14 days according to length of hospitalization.

* Intervention group: HUK (0.15 PNA) and sodium chloride injection (100ml), once per day
* Control group: placebo (0 PNA) and sodium chloride injection (100ml), once per day The total follow-up duration is 90 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Having anterior circulation AIS within 24 hours of onset.
3. The NIHSS score at enrollment is 4 to 25.
4. Receiving intravenous recombinant tissue plasminogen activator (rt-PA) or TNK-tPA, or endovascular treatment including intra-arterial thrombolysis, mechanical thrombectomy, or intravenous rt-PA /TNK-tPA bridging endovascular treatment.
5. Being independent in daily activities (mRS ≤1) before onset.
6. Patients or their legal representatives are able and willing to sign informed consent forms.

Exclusion Criteria:

1. Having an Alberta Stroke Program Early Computed Tomography Score (ASPECT) score of 6 or less confirmed by preoperational computed tomography scan.
2. Being already treated with HUK or any drugs containing HUK after onset.
3. Having an allergy history of HUK or drugs containing HUK, or other drugs and food.
4. Having a history of coagulation dysfunction, systemic bleeding, or thrombocytopenia; having hemorrhagic diseases at the time of enrollment, including cerebral hemorrhage, subarachnoid hemorrhage, epidural or subdural hematoma, gingival bleeding, gastrointestinal bleeding, dermal ecchymosis, etc; taking anticoagulants including warfarin, rivaroxaban, etc.; or taking heparin within 48 hours after stroke onset.
5. Taking angiotensin-converting enzyme inhibitor (ACEI) antihypertensive drugs regularly within one week before enrollment, including captopril, enalapril, benazepril, etc.
6. Having chronic liver disease or liver dysfunction, with elevated ALT/AST (>3.0×ULN ); or having kidney dysfunction or receiving dialysis, with elevated serum creatinine (>2.0×ULN).
7. Having severe cardiopulmonary disease that are deemed unsuitable for the study by the investigators.
8. Having contraindications for intravenous thrombolysis or endovascular treatment, including intra-arterial thrombolysis, mechanical thrombectomy, or intravenous rt-PA /TNK-tPA bridging endovascular treatment.
9. Having lethal diseases with a life expectancy < 3 months.
10. Being pregnant or lactating; or women of child-bearing age not taking effective contraception, or having no negative pregnancy test record.
11. Being unable to complete the study due to mental illness, cognitive or emotional disorder, physical condition, geographical factors, etc.
12. Participating in another clinical trial currently.
13. Other conditions that investigators consider he/she is not appropriate to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1204 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of a favorable outcome (mRS 0-2) | at 90 days
  The proportion of a favorable outcome, defined by a modified Rankin Scale (mRS) score ranging from 0 to 2, reflects the percentage of patients who attained a functional status from no symptoms to mild disability, enabling them to perform all pre-stroke activities without assistance.

SECONDARY OUTCOMES:
Proportion of a favorable outcome (mRS 0-2) | at 14 days
  The proportion of a favorable outcome, defined by a modified Rankin Scale (mRS) score ranging from 0 to 2, reflects the percentage of patients who attained a functional status from no symptoms to mild disability, enabling them to perform all pre-stroke activities without assistance.
Proportion of an excellent outcome (mRS 0-1) | at 90 days
  The proportion of an excellent outcome, characterized by a modified Rankin Scale (mRS) score of 0 to 1, represents the percentage of patients who achieved a functional status from no symptoms to no significant disability despite symptoms, allowing them to resume all pre-stroke activities without any aid.
Distribution of mRS score | at 90 days
  The distribution of modified Rankin Scale (mRS) scores provides a comprehensive overview of the functional outcomes across a patient population, categorizing the degree of disability from no symptoms (score 0) to severe disability or death (score 6).
Improvement of NIHSS score | at 14 days
  The improvement of the National Institutes of Health Stroke Scale (NIHSS) score serves as a quantifiable measure of neurological recovery, reflecting the reduction in stroke-related deficits and the enhancement of patient functional capabilities over time. Minimum Score: 0 (no stroke symptoms) Maximum Score: 42 (severe stroke) Higher NIHSS scores indicate more severe stroke symptoms and are associated with worse outcomes.Lower NIHSS scores indicate milder stroke symptoms and are associated with better outcomes.
Risk of recurrent symptomatic stroke | within 90 days
  The risk of recurrent symptomatic stroke quantifies the probability of a subsequent stroke event with clinical manifestations, providing a critical measure for assessing the long-term efficacy of stroke prevention strategies and the ongoing vulnerability of the patient population.
Risk of recurrent symptomatic ischemic stroke | within 90 days
  The risk of recurrent symptomatic ischemic stroke delineates the likelihood of a subsequent ischemic stroke event accompanied by clinical symptoms, serving as a pivotal indicator for evaluating the effectiveness of secondary prevention measures and the persistent threat of cerebral ischemia in affected individuals.
Risk of combined vascular events | within 90 days
  The risk of combined vascular events encompasses the probability of experiencing any major vascular incident, such as stroke, myocardial infarction, or vascular death, offering a comprehensive metric for assessing the overall burden of vascular disease and the aggregate impact of therapeutic interventions on cardiovascular health.
Improvement of EQ-5D-5L | at 90 days
  The improvement of EQ-5D-5L(EuroQol 5-Dimension 5-Level) reflects an enhancement in health-related quality of life, as measured by gains across five dimensions-mobility, self-care, usual activities, pain/discomfort, and anxiety/depression-on a five-level severity scale, indicating a positive shift in the patient's overall health state and well-being.
  Minimum Score: 0 (worst imaginable health state) Maximum Score: 100 (best imaginable health state) For the descriptive system, a lower score (closer to 11111) indicates better health-related quality of life, while a higher score (closer to 55555) indicates worse health-related quality of life.
  For the VAS, a higher score (closer to 100) indicates better self-rated health, while a lower score (closer to 0) indicates worse self-rated health.
Improvement of MOCA | at 90 days
  The improvement of the Montreal Cognitive Assessment (MoCA) score signifies an enhancement in cognitive function, encompassing domains such as attention, memory, language, and executive functions, thereby indicating a positive progression in the patient's cognitive status and potential recovery from cognitive impairment.
  Minimum Score: 0 (severe cognitive impairment) Maximum Score: 30 (no cognitive impairment) Higher MoCA scores indicate better cognitive function. Lower MoCA scores indicate worse cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Yilong, MD, PhD, Study Chair — Beijing Tiantan Hospital; Wang Tingting, MD, Study Director — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Y, Xu J, Zhao X, Wang D, Wang C, Liu L, Wang A, Meng X, Li H, Wang Y. Association of hypertension with stroke recurrence depends on ischemic stroke subtype. Stroke. 2013 May;44(5):1232-7. doi: 10.1161/STROKEAHA.111.000302. Epub 2013 Feb 26. PMID 23444308
- [Background] Pan Y, Li Z, Li J, Jin A, Lin J, Jing J, Li H, Meng X, Wang Y, Wang Y. Residual Risk and Its Risk Factors for Ischemic Stroke with Adherence to Guideline-Based Secondary Stroke Prevention. J Stroke. 2021 Jan;23(1):51-60. doi: 10.5853/jos.2020.03391. Epub 2021 Jan 31. PMID 33600702
- [Background] Emberson J, Lees KR, Lyden P, Blackwell L, Albers G, Bluhmki E, Brott T, Cohen G, Davis S, Donnan G, Grotta J, Howard G, Kaste M, Koga M, von Kummer R, Lansberg M, Lindley RI, Murray G, Olivot JM, Parsons M, Tilley B, Toni D, Toyoda K, Wahlgren N, Wardlaw J, Whiteley W, del Zoppo GJ, Baigent C, Sandercock P, Hacke W; Stroke Thrombolysis Trialists' Collaborative Group. Effect of treatment delay, age, and stroke severity on the effects of intravenous thrombolysis with alteplase for acute ischaemic stroke: a meta-analysis of individual patient data from randomised trials. Lancet. 2014 Nov 29;384(9958):1929-35. doi: 10.1016/S0140-6736(14)60584-5. Epub 2014 Aug 5. PMID 25106063
- [Background] Asadi H, Dowling R, Yan B, Wong S, Mitchell P. Advances in endovascular treatment of acute ischaemic stroke. Intern Med J. 2015 Aug;45(8):798-805. doi: 10.1111/imj.12652. PMID 25443686
- [Background] Berkhemer OA, Fransen PS, Beumer D, van den Berg LA, Lingsma HF, Yoo AJ, Schonewille WJ, Vos JA, Nederkoorn PJ, Wermer MJ, van Walderveen MA, Staals J, Hofmeijer J, van Oostayen JA, Lycklama a Nijeholt GJ, Boiten J, Brouwer PA, Emmer BJ, de Bruijn SF, van Dijk LC, Kappelle LJ, Lo RH, van Dijk EJ, de Vries J, de Kort PL, van Rooij WJ, van den Berg JS, van Hasselt BA, Aerden LA, Dallinga RJ, Visser MC, Bot JC, Vroomen PC, Eshghi O, Schreuder TH, Heijboer RJ, Keizer K, Tielbeek AV, den Hertog HM, Gerrits DG, van den Berg-Vos RM, Karas GB, Steyerberg EW, Flach HZ, Marquering HA, Sprengers ME, Jenniskens SF, Beenen LF, van den Berg R, Koudstaal PJ, van Zwam WH, Roos YB, van der Lugt A, van Oostenbrugge RJ, Majoie CB, Dippel DW; MR CLEAN Investigators. A randomized trial of intraarterial treatment for acute ischemic stroke. N Engl J Med. 2015 Jan 1;372(1):11-20. doi: 10.1056/NEJMoa1411587. Epub 2014 Dec 17. PMID 25517348
- [Background] Goyal M, Demchuk AM, Menon BK, Eesa M, Rempel JL, Thornton J, Roy D, Jovin TG, Willinsky RA, Sapkota BL, Dowlatshahi D, Frei DF, Kamal NR, Montanera WJ, Poppe AY, Ryckborst KJ, Silver FL, Shuaib A, Tampieri D, Williams D, Bang OY, Baxter BW, Burns PA, Choe H, Heo JH, Holmstedt CA, Jankowitz B, Kelly M, Linares G, Mandzia JL, Shankar J, Sohn SI, Swartz RH, Barber PA, Coutts SB, Smith EE, Morrish WF, Weill A, Subramaniam S, Mitha AP, Wong JH, Lowerison MW, Sajobi TT, Hill MD; ESCAPE Trial Investigators. Randomized assessment of rapid endovascular treatment of ischemic stroke. N Engl J Med. 2015 Mar 12;372(11):1019-30. doi: 10.1056/NEJMoa1414905. Epub 2015 Feb 11. PMID 25671798
- [Background] Campbell BC, Mitchell PJ, Kleinig TJ, Dewey HM, Churilov L, Yassi N, Yan B, Dowling RJ, Parsons MW, Oxley TJ, Wu TY, Brooks M, Simpson MA, Miteff F, Levi CR, Krause M, Harrington TJ, Faulder KC, Steinfort BS, Priglinger M, Ang T, Scroop R, Barber PA, McGuinness B, Wijeratne T, Phan TG, Chong W, Chandra RV, Bladin CF, Badve M, Rice H, de Villiers L, Ma H, Desmond PM, Donnan GA, Davis SM; EXTEND-IA Investigators. Endovascular therapy for ischemic stroke with perfusion-imaging selection. N Engl J Med. 2015 Mar 12;372(11):1009-18. doi: 10.1056/NEJMoa1414792. Epub 2015 Feb 11. PMID 25671797
- [Background] Saver JL, Goyal M, Bonafe A, Diener HC, Levy EI, Pereira VM, Albers GW, Cognard C, Cohen DJ, Hacke W, Jansen O, Jovin TG, Mattle HP, Nogueira RG, Siddiqui AH, Yavagal DR, Baxter BW, Devlin TG, Lopes DK, Reddy VK, du Mesnil de Rochemont R, Singer OC, Jahan R; SWIFT PRIME Investigators. Stent-retriever thrombectomy after intravenous t-PA vs. t-PA alone in stroke. N Engl J Med. 2015 Jun 11;372(24):2285-95. doi: 10.1056/NEJMoa1415061. Epub 2015 Apr 17. PMID 25882376
- [Background] Zi W, Qiu Z, Li F, Sang H, Wu D, Luo W, Liu S, Yuan J, Song J, Shi Z, Huang W, Zhang M, Liu W, Guo Z, Qiu T, Shi Q, Zhou P, Wang L, Fu X, Liu S, Yang S, Zhang S, Zhou Z, Huang X, Wang Y, Luo J, Bai Y, Zhang M, Wu Y, Zeng G, Wan Y, Wen C, Wen H, Ling W, Chen Z, Peng M, Ai Z, Guo F, Li H, Guo J, Guan H, Wang Z, Liu Y, Pu J, Wang Z, Liu H, Chen L, Huang J, Yang G, Gong Z, Shuai J, Nogueira RG, Yang Q; DEVT Trial Investigators. Effect of Endovascular Treatment Alone vs Intravenous Alteplase Plus Endovascular Treatment on Functional Independence in Patients With Acute Ischemic Stroke: The DEVT Randomized Clinical Trial. JAMA. 2021 Jan 19;325(3):234-243. doi: 10.1001/jama.2020.23523. PMID 33464335
- [Background] Yang P, Zhang Y, Zhang L, Zhang Y, Treurniet KM, Chen W, Peng Y, Han H, Wang J, Wang S, Yin C, Liu S, Wang P, Fang Q, Shi H, Yang J, Wen C, Li C, Jiang C, Sun J, Yue X, Lou M, Zhang M, Shu H, Sun D, Liang H, Li T, Guo F, Ke K, Yuan H, Wang G, Yang W, Shi H, Li T, Li Z, Xing P, Zhang P, Zhou Y, Wang H, Xu Y, Huang Q, Wu T, Zhao R, Li Q, Fang Y, Wang L, Lu J, Li Y, Fu J, Zhong X, Wang Y, Wang L, Goyal M, Dippel DWJ, Hong B, Deng B, Roos YBWEM, Majoie CBLM, Liu J; DIRECT-MT Investigators. Endovascular Thrombectomy with or without Intravenous Alteplase in Acute Stroke. N Engl J Med. 2020 May 21;382(21):1981-1993. doi: 10.1056/NEJMoa2001123. Epub 2020 May 6. PMID 32374959
- [Background] Wang H, Zi W, Hao Y, Yang D, Shi Z, Lin M, Wang S, Liu W, Wang Z, Liu X, Guo F, Liu Y, Xu G, Xiong Y, Liu X; ACTUAL Investigators. Direct endovascular treatment: an alternative for bridging therapy in anterior circulation large-vessel occlusion stroke. Eur J Neurol. 2017 Jul;24(7):935-943. doi: 10.1111/ene.13311. Epub 2017 May 11. PMID 28493511
- [Background] Ye Q, Zhai F, Chao B, Cao L, Xu Y, Zhang P, Han H, Wang L, Xu B, Chen W, Wen C, Wang S, Wang R, Zhang L, Jiao L, Liu S, Zhu YC, Wang LD. Rates of intravenous thrombolysis and endovascular therapy for acute ischaemic stroke in China between 2019 and 2020. Lancet Reg Health West Pac. 2022 Feb 22;21:100406. doi: 10.1016/j.lanwpc.2022.100406. eCollection 2022 Apr. PMID 35243459
- [Background] Shen H, Killingsworth MC, Bhaskar SMM. Comprehensive Meta-Analysis of Futile Recanalization in Acute Ischemic Stroke Patients Undergoing Endovascular Thrombectomy: Prevalence, Factors, and Clinical Outcomes. Life (Basel). 2023 Sep 26;13(10):1965. doi: 10.3390/life13101965. PMID 37895347
- [Background] Wang A, Jia B, Zhang X, Huo X, Chen J, Gui L, Cai Y, Guo Z, Han Y, Peng Z, Jing P, Chen Y, Liu Y, Yang Y, Wang F, Sun Z, Li T, Sun H, Yuan H, Shao H, Gao L, Zhang P, Wang F, Cao X, Shi W, Li C, Yang J, Zhang H, Wang F, Deng J, Liu Y, Deng W, Song C, Chen H, He L, Zhao H, Li X, Yang H, Zhou Z, Wang Y, Miao Z; BAST Investigators. Efficacy and Safety of Butylphthalide in Patients With Acute Ischemic Stroke: A Randomized Clinical Trial. JAMA Neurol. 2023 Aug 1;80(8):851-859. doi: 10.1001/jamaneurol.2023.1871. PMID 37358859
- [Background] Ling L, Hou Q, Xing S, Yu J, Pei Z, Zeng J. Exogenous kallikrein enhances neurogenesis and angiogenesis in the subventricular zone and the peri-infarction region and improves neurological function after focal cortical infarction in hypertensive rats. Brain Res. 2008 Apr 24;1206:89-97. doi: 10.1016/j.brainres.2008.01.099. Epub 2008 Mar 19. PMID 18353282
- [Background] Xia CF, Yin H, Yao YY, Borlongan CV, Chao L, Chao J. Kallikrein protects against ischemic stroke by inhibiting apoptosis and inflammation and promoting angiogenesis and neurogenesis. Hum Gene Ther. 2006 Feb;17(2):206-19. doi: 10.1089/hum.2006.17.206. PMID 16454654
- [Background] Miao J, Deng F, Zhang Y, Xie HY, Feng JC. Exogenous human urinary kallidinogenase increases cerebral blood flow in patients with acute ischemic stroke. Neurosciences (Riyadh). 2016 Apr;21(2):126-30. doi: 10.17712/nsj.2016.2.20150581. PMID 27094522
- [Background] Li J, Chen Y, Zhang X, Zhang B, Zhang M, Xu Y. Human Urinary Kallidinogenase Improves Outcome of Stroke Patients by Shortening Mean Transit Time of Perfusion Magnetic Resonance Imaging. J Stroke Cerebrovasc Dis. 2015 Aug;24(8):1730-7. doi: 10.1016/j.jstrokecerebrovasdis.2015.03.032. Epub 2015 Jun 29. PMID 26139453
- [Background] Zhang C, Tao W, Liu M, Wang D. Efficacy and safety of human urinary kallidinogenase injection for acute ischemic stroke: a systematic review. J Evid Based Med. 2012 Feb;5(1):31-9. doi: 10.1111/j.1756-5391.2012.01167.x. PMID 23528118
- [Background] Huang Y, Wang B, Zhang Y, Wang P, Zhang X. Efficacy and safety of human urinary kallidinogenase for acute ischemic stroke: a meta-analysis. J Int Med Res. 2020 Sep;48(9):300060520943452. doi: 10.1177/0300060520943452. PMID 32954870
- [Background] Wang YD, Lu RY, Huang XX, Yuan F, Hu T, Peng Y, Huang SQ. Human tissue kallikrein promoted activation of the ipsilesional sensorimotor cortex after acute cerebral infarction. Eur Neurol. 2011;65(4):208-14. doi: 10.1159/000325735. Epub 2011 Mar 22. PMID 21422759
- [Background] Yan X, Chen H, Shang X. Human urinary kallidinogenase decreases the incidence of post-stroke cognitive impairment in acute ischemic stroke patients. J Integr Neurosci. 2022 Apr 8;21(3):80. doi: 10.31083/j.jin2103080. PMID 35633161
- [Background] Han D, Chen X, Li D, Liu S, Lyu Y, Feng J. Human Urinary Kallidinogenase decreases recurrence risk and promotes good recovery. Brain Behav. 2018 Aug;8(8):e01033. doi: 10.1002/brb3.1033. Epub 2018 Jul 20. PMID 30030910
- [Background] Wu J, Wu J, Wang L, Liu J. Urinary Kallidinogenase plus rt-PA Intravenous Thrombolysis for Acute Ischemic Stroke: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Comput Math Methods Med. 2022 May 17;2022:1500669. doi: 10.1155/2022/1500669. eCollection 2022. PMID 35620206